CLINICAL TRIAL: NCT05465005
Title: Perception of Electrical Stimuli During Muscle Activation in Individuals with Stroke
Brief Title: Perception of Electrical Stimuli in Individuals with Stroke
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Netta Gurari (Other)
Collaborators: Northwestern University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Virginia Polytechnic Institute and State University (Other)
Responsible Party: Sponsor-Investigator, Netta Gurari, Assistant Professor, Virginia Polytechnic Institute and State University
Organization: Virginia Polytechnic Institute and State University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: K25HD096116 (NIH); K25HD096116 (NIH)
Record Dates: First submitted 2022-07-15; First posted 2022-07-19 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Stroke
Keywords: tactile perception; somatosensation; muscle activation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: We will compare outcome measures across three experimental conditions and each upper extremity in participants with stroke and similarly-aged controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Behavioral: Torque Generation — Relaxed, or flexing about the elbow to 25% or 50% of the maximum elbow torque that one can generate.
  Other Names: Muscle activation

SUMMARY:
To successfully manipulate objects in one's surroundings, such as when lifting a cup, one must accurately perceive their physical interactions. This includes accurately interpreting the tactile cues arising at one's fingertips when touching an object. Currently, tactile perception is assessed in individuals with stroke using passive protocols. Research has yet to explore whether activating one's muscles impacts the tactile perceptual process in individuals with stroke despite previous research demonstrating the effect of muscle activation on tactile perception in individuals who are neurologically intact. The proposed research will be the first to address the impact of muscle activation, in addition to stroke, on tactile perception. As such, the proposed research is significant for advancing our understanding of the extent to which tactile deficits occur in individuals with stroke, particularly during volitional movement.

DETAILED DESCRIPTION:
Participants will detect an externally-applied electrical stimulus at their fingertip with the elbow: 1) relaxed and flexed to 2) 25% and 3) 50% of their maximum voluntary torque (MVT). We will compare the detection threshold for these three conditions between each arm of participants with stroke and similarly-aged controls. Based on pilot data, we hypothesize that the detection threshold will be largest at the paretic arm when flexing to 50% MVT due to the greatest inhibition of sensory signals. Findings will indicate whether stroke negatively impacts an individual's ability to detect tactile stimuli during volitional sensorimotor tasks.

ELIGIBILITY:
Inclusion Criteria:

* For the participants with stroke, i) a single unilateral cortical lesion that took place at least one year prior and ii) an absence of comorbid neurological impairments
* Ability to understand and complete the experimental tasks
* Capacity to provide informed consent
* At least 18 years of age

Exclusion Criteria:

* Major injury to either arm
* Sensory neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Detection threshold | ~5 minutes
  Minimum magnitude of current at which an electrical stimulus can be detected

CONTACTS AND LOCATIONS:
Locations (1):
- Virginia Tech Biomedical Engineering and Mechanics, Blacksburg, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Post LJ, Zompa IC, Chapman CE. Perception of vibrotactile stimuli during motor activity in human subjects. Exp Brain Res. 1994;100(1):107-20. doi: 10.1007/BF00227283. PMID 7813639
- [Background] Chapman, C. E., Zompa, I. C., Williams, S. R., Shenasa, J. & Jiang, W. Factors influencing the perception of tactile stimuli during movement. in Somesthesis and the Neurobiology of the Somatosensory Cortex (eds. Franzén, O., Johansson, R. & Terenius, L.) 307-320 (Birkhäuser Basel, 1996).
- [Background] Seki K, Perlmutter SI, Fetz EE. Sensory input to primate spinal cord is presynaptically inhibited during voluntary movement. Nat Neurosci. 2003 Dec;6(12):1309-16. doi: 10.1038/nn1154. Epub 2003 Nov 16. PMID 14625555
- [Background] Pavlenko, V. B. Self-initiated motor behavioral act-related neuronal activity in the cat Locus Coeruleus. Neurophysiology 35, 29-37 (2003).
- [Background] Wei K, Glaser JI, Deng L, Thompson CK, Stevenson IH, Wang Q, Hornby TG, Heckman CJ, Kording KP. Serotonin affects movement gain control in the spinal cord. J Neurosci. 2014 Sep 17;34(38):12690-700. doi: 10.1523/JNEUROSCI.1855-14.2014. PMID 25232107
- [Background] Jacobs BL, Martin-Cora FJ, Fornal CA. Activity of medullary serotonergic neurons in freely moving animals. Brain Res Brain Res Rev. 2002 Oct;40(1-3):45-52. doi: 10.1016/s0165-0173(02)00187-x. PMID 12589905
- [Background] Seki K, Fetz EE. Gating of sensory input at spinal and cortical levels during preparation and execution of voluntary movement. J Neurosci. 2012 Jan 18;32(3):890-902. doi: 10.1523/JNEUROSCI.4958-11.2012. PMID 22262887